CLINICAL TRIAL: NCT00002750
Title: Phase I of Intrathecal Melphalan in Patients With Recurrent Neoplastic Meningitis
Brief Title: Melphalan in Patients With Neoplastic Meningitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 2117; DUMC-2117-00-11R8; DUMC-1631-96-11R4; DUMC-1728-97-11R5; DUMC-1818-98-11R6; DUMC-1961-99-11R7; NCI-V96-0869; CDR0000064684 (Other: NCI)
Record Dates: First submitted 1999-11-01; First posted 2004-05-24 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Brain and Central Nervous System Tumors; Extragonadal Germ Cell Tumor; Leukemia; Lymphoma; Ovarian Cancer
Keywords: recurrent childhood acute lymphoblastic leukemia; recurrent adult Hodgkin lymphoma; Waldenström macroglobulinemia; recurrent childhood lymphoblastic lymphoma; childhood central nervous system germ cell tumor; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; recurrent/refractory childhood Hodgkin lymphoma; recurrent ovarian germ cell tumor; recurrent adult non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; extragonadal germ cell tumor; leptomeningeal metastases; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Leukemia; Lymphoma; Ovarian Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Hodgkin Disease; Waldenstrom Macroglobulinemia; Leukemia, Myeloid, Acute; Recurrence; Lymphoma, Non-Hodgkin; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Meningeal Carcinomatosis; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Melphalan

INTERVENTIONS:
Drug: melphalan

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of melphalan in patients with persistent or recurrent neoplastic meningitis.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of intrathecal melphalan (L-PAM) in patients with neoplastic meningitis. II. Determine the CSF and serum pharmacokinetics of L-PAM administered via an Ommaya reservoir to these patients.

OUTLINE: This is a dose escalation study. Patients receive melphalan (L-PAM) intrathecally (IT) via lumbar puncture or Ommaya reservoir twice a week for 2 weeks. Cohorts of 3-6 patients receive escalating doses of melphalan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 4 of 6 patients experience dose-limiting toxicity. At least 3 patients receive L-PAM via Ommaya reservoir at the MTD. Patients with objective or significant clinical response may receive additional L-PAM IT once a week for 2 consecutive weeks, every other week for 2 doses, and then monthly thereafter. Patients are followed every 12 weeks for 1 year or until disease progression.

PROJECTED ACCRUAL: A minimum of 3 children and 3 adults per dose level will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed malignancy that is metastatic to the CSF or leptomeningeal/subarachnoid space, including the following: Leukemia Lymphoma Germ cell tumors Persistent or recurrent disease required Cytologic evidence of malignancy in CSF or evidence of leptomeningeal tumor by CT or MRI No obstructive hydrocephalus or complete block of spinal CSF pathways on pre- study MRI or CT No rapidly progressing or deteriorating neurological deficit

PATIENT CHARACTERISTICS: Age: 3 and over Performance status: Karnofsky 60-100% (age 10 and over) OR Lansky 60-100% (age under 10) Life expectancy: At least 8 weeks Hematopoietic: Absolute neutrophil count greater than 1,000/mm3* Platelet count greater than 100,000/mm3* * Lower values allowed with approval of the investigator Hepatic: Bilirubin less than 3.0 mg/dL Renal: Creatinine less than 2 mg/dL Blood urea nitrogen less than 30 mg/dL Electrolytes (including calcium, magnesium, phosphate) normal Other: No active infection Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Prior systemic chemotherapy within 3 weeks of entry allowed at investigator's discretion At least 3 weeks since prior intrathecal chemotherapy No other concurrent intrathecal chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 3 weeks since prior radiotherapy to the CNS No concurrent radiotherapy to the CNS Surgery: Not specified

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 1992-12; Primary Completion 2001-05 (Actual); Study Completion 2001-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry S. Friedman, MD, Study Chair — Duke Cancer Institute
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States